CLINICAL TRIAL: NCT02037139
Title: Primary Care Intervention Promoting Hearing Health Care Service Access and Use
Brief Title: Hearing Health Care Service Access and Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 4R33DC011510-03 (NIH)
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Hearing Loss
Keywords: Hearing loss; Screening; Primary Care
MeSH Terms: conditions — Hearing Loss | interventions — Mass Screening; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (screening) (Active Comparator): screening only (standard care control)
  Interventions: Other: Screening
- Educational brochure (Active Comparator): Screening + illustrated educational brochure
  Interventions: Other: Screening; Other: Brochure
- Education (Experimental): Screening + illustrated educational brochure + an in-person educational intervention
  Interventions: Other: Screening; Other: Brochure; Behavioral: Education

INTERVENTIONS:
Other: Screening — Standard care screening
Other: Brochure — Participants are given an illustrated educational brochure
  Arms: Education; Educational brochure
Behavioral: Education — Participants undergo a in-person educational intervention
  Arms: Education

SUMMARY:
Hearing loss screening rates in for older persons in primary care clinics are very low even though hearing loss is relatively common for older persons. When diagnosed with hearing loss older persons are often reluctant to follow through. This study involves a prospective controlled trial comparing the effectiveness of three primary care based protocols for older adults ≥ 60 who screen positive for possible hearing loss in promoting subsequent access to and use of hearing health care services. The protocols will compare: 1) screening only (standard care control); 2) screening plus an illustrated educational brochure; and 3) screening plus an in-person educational intervention and an illustrated educational brochure. Screening will be done by primary care personnel. Participants will be tracked for 8 months to assess outcomes.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the extent to which hearing health outcomes are improved when patients are screened for hearing loss and provided an educational brochure or screened and provided the brochure plus an educational segment emphasizing points in the brochure versus a standard screening only protocol. These procedures are non-invasive. Hearing loss screening is part of basic health evaluations for older persons, brochures are commonly handed out for a variety of health conditions, and providing patient education is common practice.

At all sites our study research nurse will train clinic staff, contact patients who have indicated they are interested in taking part, obtain informed consent, administer baseline and follow-up questionnaires, and ensure that those completing the two follow-ups receive their gift cards. No information from clinic medical records will be obtained.

Aims:

1. Evaluate the extent to which hearing health outcomes are improved when patients are screened for hearing loss and provided an educational brochure or screened and provided the brochure plus an educational segment emphasizing points in the brochure versus a standard screening only protocol..
2. Examine hearing health outcomes by patient and clinic characteristics.
3. Compare any observed gains in outcomes against the estimated staff time to administer either the brochure or the brochure plus the educational segment.

The three primary outcomes involve comparing the differential impacts of adding an illustrated educational brochure or adding both a brochure and a brief educational segment over screening only. These three outcomes are whether the participant went to see a hearing specialist for an evaluation, whether a hearing or other assistive listening device was obtained if recommended, and whether the device if obtained was being used. Other outcomes include the number of hours a day participants who received assistive devices actually wear them, the number of changes participants have made to improve communication other than obtaining an assistive device, and the extent to which their hearing related quality of life improves.

The primary care clinics taking part in our study already do some screening for hearing loss but often screening is not perceived as leading to better outcomes. The clinics are interested in the opportunity to participate in a project that will assess how effective screening is when combined with additional educational material. All consenting and data collection will be done by our study's Research Nurse.

Specific procedures are:

1. Older patients coming into the clinic for a medical appointment and who are not wearing hearing aids will be screened by intake personnel (usually a medical assistant or office nurse) for hearing loss using a direct question ("Do you have any difficulty hearing?") and a finger rub test (the finger rub protocol is attached). When either or both of these tests indicate possible hearing loss, intake personnel will tell the patient that their health care provider will be informed and then ask them if they are interested in taking part in a study of hearing loss. Those who express an interest will be asked to fill out contact information on a card for transmission to the study's Research Nurse. They will also be given a flyer describing the study and two copies of the consent to take with them to review and discuss with the study's research nurse. A stamped return envelope will be included for mailing the signed consent after discussing the study with the Research Nurse. The envelope will have the study address both on the front and in the space for the return address in order to protect patient confidentiality.

   One of three protocols will then occur for those indicating an interest in the study:
   * For the first 28 patients the intake personnel will take no further action other than to provide the screening results to the patient's health care provider.
   * For the next 28 patients the intake personnel will hand them the brochure For the last 28 patients the intake personnel will hand them the brochure and then ask if it is all right with them if he/she goes over some points in the brochure.
2. Training for the finger rub and what to do during the three protocols will be conducted by the study's Research Nurse.
3. The health care provider that the patient sees will follow his or her usual procedures for handling a patient with possible hearing loss. This usually involves checking the ears for wax buildup, further discussion about the possible extent of the loss, and referral to a hearing specialist if warranted.
4. The Research Nurse will come by the clinics regularly to pick up the contact cards and respond to any questions that medical assistants or other clinic staff may have.
5. The Research Nurse will then contact potential participants to explain the study, review the consent they took home, ask those still interested in taking part in the study to sign one copy of the consent and place it in the provided envelope for mailing, and administer the baseline questionnaire. She will explain that there will be two follow-up contacts at 4 and 8 months. If participants can hear well enough to do the interviewing over the telephone it will be used for all contact between the Research Nurse and participants. The informed consent will include a self-addressed envelope for mailing the signed copy to the Research Nurse. If participants do not feel they can hear well enough to talk with the Research Nurse over the telephone, all consenting and interviewing will be done at a place of their own choosing.
6. At the end of the 8-month follow-up, participants from the first two protocol groups will be given the same educational materials (brochure and/or verbal educational protocol) by the study Research Nurse that they would have received had they been in the third protocol group. Thus by the end of the study all participants will have received the brochure and the educational intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older
* Not currently wearing a hearing aid
* Cognitively capable of giving informed consent
* Able to speak and understand English
* No concurrent health problem that would limit participation
* Screen positive for hearing loss using single question and/or finger rub

Exclusion Criteria:

* Age 59 or less
* Currently wearing a hearing aid
* Cognitively impaired or not cognitively capable of giving informed consent
* Unable to speak and understand English
* Has a concurrent health condition that limits participation
* Does not screen positive for hearing loss

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Referral rates for hearing evaluation | 8 months after initial screening
  Proportion of those who screened positive for possible hearing loss who follow through on clinic recommendations for referrals or who elect a referral on their own

SECONDARY OUTCOMES:
Number of changes made to improve hearing | 8 months after initial screening
  Other than adopting hearing aids, how many changes did participants make to improve their hearing since screened. Education segment lists 6 possible changes.

OTHER OUTCOMES:
Hearing outcomes | 8 months following initial screening
  Improvement in hearing over the course of the study as assessed by the Hearing Handicap Inventory for the Elderly (HHIE-S) and Inner Ear scales

CONTACTS AND LOCATIONS:
Overall Officials: Margaret I Wallhagen, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No